CLINICAL TRIAL: NCT02907099
Title: A Phase IIb Pilot Study to Assess the Efficacy, Safety, and Pharmacodynamics Effects of Pembrolizumab and BL-8040 in Patients With Metastatic Pancreatic Cancer
Brief Title: Pembrolizumab and CXCR4 Antagonist BL-8040 in Treating Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0410; NCI-2016-01956 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0410 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-09-13; First posted 2016-09-20 (Estimated); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; Recurrent Pancreatic Adenocarcinoma; Stage IV Pancreatic Cancer AJCC v6 and v7
MeSH Terms: interventions — 4-fluorobenzoyl-TN-14003; BKT140; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CXCR4 antagonist BL-8040, pembrolizumab) (Experimental): Patients receive CXCR4 antagonist BL-8040 SC on days 1-5 and 8-12 of cycle 1 and days 1, 4, 8, and 11 of subsequent cycles. Beginning cycle 2, patients also receive pembrolizumab IV over about 30 minutes on day 1. Cycles repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: CXCR4 Antagonist BL-8040; Biological: Pembrolizumab; Other: Pharmacological Study

INTERVENTIONS:
Drug: CXCR4 Antagonist BL-8040 — Given SC
  Other Names: BKT140; BL-8040
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Pharmacological Study — Correlative studies

SUMMARY:
This pilot phase IIb trial studies how well pembrolizumab and CXCR4 antagonist BL-8040 work in treating patients with pancreatic cancer that has spread to other places. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. CXCR4 antagonist BL-8040 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving pembrolizumab and CXCR4 antagonist BL-8040 may work better in treating patients with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the overall response rate (complete response or partial response) after treatment with CXCR4 antagonist BL-8040 (BL-8040) and pembrolizumab.

SECONDARY OBJECTIVES:

I. To determine the ability of BL-8040 by itself and in combination with pembrolizumab to increase T cell infiltration into the tumor.

II. To determine if BL-8040 treatment results in increases in circulating immune cells.

III. To estimate the safety and tolerability of intravenous administration of pembrolizumab in combination with sub-cutaneously injected BL-8040 in subjects with advanced pancreatic cancer.

EXPLORATORY OBJECTIVES:

I. To evaluate overall response rate (ORR) per immune-related (ir) Response Evaluation Criteria in Solid Tumors (RECIST) and duration of response (DOR), disease control rate (DCR), time to progression (TTP), progression free survival (PFS), and overall survival (OS) per RECIST and irRECIST assessed by MD Anderson investigators.

II. To explore the association between PD-L1 expression by immunohistochemistry, shed PD-L1 level, somatic gene expression profiling and antitumor efficacy of pembrolizumab based on RECIST 1.1 imaging criteria as well as overall survival.

III. To explore the relationship between genomic variation and response to the treatment administered.

IV. Tissue and blood immune monitoring will be conducted through our immune platform group as detailed per the biomarker section based on 3 biopsies done at the following time points: 1) pre-treatment, 2) during the third week of cycle 2 or beginning of cycle 3, and 3) voluntary upon end of cycle 1 (BL-8040 [BL] monotherapy) on days 10 to 14.

OUTLINE:

Patients receive CXCR4 antagonist BL-8040 subcutaneously (SC) on days 1-5 and 8-12 of cycle 1 and days 1, 4, 8, and 11 of subsequent cycles. Beginning cycle 2, patients also receive pembrolizumab intravenously (IV) over about 30 minutes on day 1. Cycles repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 10 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma based on pathology report
* Be willing and able to provide written informed consent for the trial
* Have measurable disease based on RECIST 1.1; target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Have documented objective radiographic progression after stopping treatment with first-line therapy; Note: the same image acquisition and processing parameters should be used throughout the study for a given subject
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion from a metastatic site; newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on day 1; subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from Merck; the specimen must be from a biopsy site that would be accessible for at least one subsequent biopsy after initiation on the trial
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Have a predicted life expectancy of greater than 3 months
* Absolute neutrophil count (ANC) >= 1,000 /mcL (performed within 10 days of treatment initiation)
* Platelets >=100,000 /mcL (performed within 10 days of treatment initiation)
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 14 days of assessment) (performed within 10 days of treatment initiation)
* Serum creatinine OR measured or calculated creatinine clearance (should be calculated per institutional standard) (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) =< 1.5 X upper limit of normal (ULN) OR >= 60 mL/min for subject with creatinine levels =< 1.5 X institutional ULN (performed within 10 days of treatment initiation)
* Serum total bilirubin =< ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > ULN (performed within 10 days of treatment initiation)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) =< 1.5 X ULN (performed within 10 days of treatment initiation)
* Albumin >= 3.3 mg/dL in the absence of dehydration (performed within 10 days of treatment initiation)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (performed within 10 days of treatment initiation)
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (performed within 10 days of treatment initiation)
* Have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication (cycle 1, day 1) (female subjects of childbearing potential); if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential must be willing to use an adequate method of contraception; contraception, for the course of the trial through 120 days after the last dose of trial drug; note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject; male subjects of childbearing potential must agree to use an adequate method of contraception; contraception, starting with the first dose of trial therapy through 120 days after the last dose of trial therapy

Exclusion Criteria:

* Has pancreatic tumor other than adenocarcinoma, including: acinar cell carcinoma, pancreaticoblastoma, malignant cystic neoplasms, endocrine neoplasms, squamous cell carcinoma; vater and periampullary duodenal or common bile duct malignancies
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy, herbal/complementary oral or IV medicine, or used an investigation device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Had a solid organ or hematologic transplant
* Has active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a diagnosed additional malignancy within 1 year prior to first dose of study treatment with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or curatively resected in situ cervical and/or breast cancers
* Has radiographically detectable (even if asymptomatic and/or previously treated) central nervous system (CNS) metastases and/or carcinomatous meningitis as assessed by principal investigator (PI) and radiology review
* Subjects excluded if there is a history of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease, or active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator, including dialysis
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment
* Has received prior immunotherapy with agents that target PD-1, PD-L1, PD-L2, CTLA-4, OX-40, or CD-137 agents, or if the subject has previously participated in Merck pembrolizumab clinical trials
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known hepatitis B or hepatitis C
* Has received a live vaccine within 30 days of planned start of study therapy (cycle 1, day 1); Note: the killed virus vaccines used for seasonal influenza vaccines for injection are allowed; however intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed
* Has a known history of active TB (Bacillus tuberculosis)
* Unable to tolerate a contrast enhanced computed tomography (CT) or magnetic resonance imaging (MRI) for staging/restaging purposes
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to such agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered small molecule agent; a. Note: subjects with =< grade 2 neuropathy or alopecia are an exception to this criterion and may qualify for the study; b. Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Patients requiring beta blockade are disqualified from participating in this study
* Patients who, in the estimation of the treating physician or primary investigator, have had a clinical deterioration of their ECOG performance within the month prior to enrollment
* The use of natural or synthetic cannabinoids
* Patients with unstable angina, new onset angina within the last 3 months, myocardial infarction within the last 6 months, and current congestive heart failure New York Heart Association class III or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon G. Smaglo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: UT Md Anderson Cancer Center
Groups:
- Pembrolizumab Plus BL-8040: In cycle 1, BL8040 was administered1.25 mg/kg s.c. daily on days 1-5 and days 8-12. Starting with the second cycle pembrolizumab was administered on day1 (200 mg) and BL8040 was continued on days 1,4,8, and 11.
  Biopsy: Pretreatment biopsies; An optional biopsy after cycle 1 (BL monotherapy) and a second mandatory biopsy after cycle 3.
Period: Overall Study
Arm/Group | Pembrolizumab Plus BL-8040
Started | 20
Completed | 15
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Not completed — Screen Fail | 2

BASELINE CHARACTERISTICS:
Population: Metastatic Pancreatic Cancer (mPC).
Arm/Group | Pembrolizumab Plus BL-8040
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 66 [23 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: To assess the overall response rate (complete response or partial response) PER RECIST 1.0 after treatment with CXCR4 antagonist BL-8040 (BL-8040) and pembrolizumab
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Plus BL-8040
Number analyzed (Participants) | 15
Participants | 1

2. Secondary Outcome: Quantity of T-Cell Infiltration Pre-treatment and Post Treatment Following Administration of BL-8040 by Itself and BL-8040 With Pembrolizumab
Description: Biomarker Analysis (TCR analysis, flow cytometry panel) of biopsy core samples was utilized to detect the presence and amount of T Cell infiltration into the tumor tissue.
Time Frame: pre treatment at baseline and post treatment (2 months)
Population: Metastatic Pancreatic Cancer (mPC)
Measure: Median (Full Range); unit: T-cells/mm^2
Arm/Group | Pembrolizumab Plus BL-8040
Number analyzed (Participants) | 6
T-cells/mm^2
  PRE TREATMENT | 52.5 [7 to 620]
  POST TREATMENT | 112.5 [20 to 420]
Statistical Analysis 1: Comparison: Pembrolizumab Plus BL-8040; Test type: Other; p = 0.5, t-test, 2 sided

3. Secondary Outcome: Quantity of Circulating T-Cells Pre-treatment and Post Treatment Following Administration of BL-8040
Description: Biomarker Analysis (TCR analysis, flow cytometry panel) of biopsy core samples was utilized to detect the Quantity of circulating T-Cells into the tumor tissue.
Time Frame: pre treatment and post treatment, up to 3 years
Measure: Median (Full Range); unit: T-cells/mm^2
Arm/Group | Pembrolizumab Plus BL-8040
Number analyzed (Participants) | 6
T-cells/mm^2
  PRE TREATMENT | 275 [100 to 2550]
  POST TREATMENT | 450 [150 to 650]
Statistical Analysis 1: Comparison: Pembrolizumab Plus BL-8040; Test type: Other; p = 0.5, t-test, 2 sided

4. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Description: Utilizing CTCAE v4.0, the number of treatment-related adverse events was recorded.
Time Frame: 2 years
Population: Metastatic Pancreatic Cancer (mPC).
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Plus BL-8040
Number analyzed (Participants) | 15
Participants | 9

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Pembrolizumab Plus BL-8040
All-Cause Mortality (participants affected / at risk) | 2/15
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 5/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab Plus BL-8040 (N=15)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hypertension (Vascular disorders) | 1
Alkaline Phosphatase increased (Investigations) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab Plus BL-8040 (N=15)
Hypertension (Vascular disorders) | 1
Alkaline Phosphatase Increased (Investigations) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Dyspnea (General disorders) | 2
Abdominal Pain (Endocrine disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT02907099/Prot_SAP_000.pdf